CLINICAL TRIAL: NCT06726824
Title: NEOnatal Multiexposure to Medical Devices Plasticizers: Endocrine Disruption MIXture Effects and Neurodevelopmental Disorders
Acronym: NEOMIX WP3
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2024 BERNARD
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Neurodevelopmental Disorder (Diagnosis)
Keywords: Neurodevelopmental disorder; Multiexposure; Medical devices; Plasticizers; Cocktail effects
MeSH Terms: conditions — Neurodevelopmental Disorders; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NEOMIX-WP3 cohort: NEOMIX-WP3 cohort corresponds to the patients incluses in the ARMED NEO cohort (NICU patients) between February 2018 And June 2019. These children are now between 6 And 7. Their parents will be asked by validated questionnaries to evaluate the Neurodevelopmental status And eventual risk factors since they got back home after NICU stay

SUMMARY:
The goal of this observational study is to evaluate the neurodevelopment of children from the ARMED NEO cohort through the ASQ3 score.

Dose the multiexposure to medical devices plasticizers during the neonatal intensive care unit stay increases the risk of developing neurodevelopmental disorders ? Patients (their parents) will complète several questionnaires (ASQ3, environnemental survey, EPICES score) during a planned teleconsultation with the research team

ELIGIBILITY:
Inclusion Criteria:

* Live patient who participated in the ARMED NEO study, included at the Clermont-Ferrand or Lille hospitals
* Patient whose holders of parental authority have expressed their non-opposition to their participation in the study

Exclusion Criteria:

* Patient whose guardians have expressed opposition to their participation in the study
* Patient with no French speaking parent
* patient

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruted in Clermont-Ferrand And Lille centers. They are ambulatory patients whose parents Will be contacted by phone by research team to plan, if they accept to participate, a teleconsultation
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ASQ3® score translated into an overall numerical score corresponding to the total of 5 dimensions of the ASQ3 test. | From enrollment to the end of the teleconsultation
ASQ3® score translated into an overall numerical score corresponding to the total of 5 dimensions of the ASQ3 test. | From en recollement to the end of the teleconsultation

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU de Lille, Lille

IPD SHARING:
Plan to Share IPD: No